CLINICAL TRIAL: NCT05459584
Title: RObotic Assisted Rehabilitation for Balance and Gait in Orthopedic Patients: Effects on Functional, Motor, and Cognitive Outcomes.
Brief Title: Robotic Assisted Rehabilitation for Balance and Gait in Orthopedic Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, GIOVANNINI SILVIA, Researcher, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0022215/22
Record Dates: First submitted 2022-07-13; First posted 2022-07-15 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis, Hip; Gait Disorders in Old Age; Balance; Distorted
Keywords: Rehabilitation; Technology; Balance
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip

STUDY DESIGN:
Intervention Model Description: Interventional pilot randomized controlled trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Technological Group (Experimental): Technological group (TG) patients will undergo robotic treatment for the improvement balance through the robotic platform (Hunova® Movendo Technology srl, Genova, IT), 3 times per week for 45 minutes each, in addition to the conventional treatment (total 180 minutes per day). In particular, the technological rehabilitation performed employing a footboard will be mostly aimed at improving the balance both in sitting and standing position, and will be proposed static and dynamic exercises, exercises dual-task exercises, and exercises to improve trunk control.
  Interventions: Device: Technological Rehabilitation
- No Intervention: Control Group (No Intervention): Congrol Group (CG) patients will undergo conventional rehabilitation treatment only, using the main rehabilitation methods (e.g., neurocognitive theory, Bobath Concept, Progressive neuromuscular facilitation, etc.).

INTERVENTIONS:
Device: Technological Rehabilitation — Specific rehabilitation for balance disorder using the robotic platform
  Other Names: Hunova® Movendo Technology srl
  Arms: Experimental: Technological Group

SUMMARY:
Osteoarthritis is a chronic, degenerative disease affecting the joints. It is characterized by the presence of bone tissue that goes to make up for the loss of articular cartilage, causing pain and limitation of movement. Osteoarthritis is a direct consequence of aging: it affects almost all 70-year-olds, peaking between 75 and 79 years. The presence of osteoarthritic processes at the hip and knee joints can result in pain, difficulty maintaining standing for a long time, and difficulty walking with loss of balance, increasing the risk of accidental falls to the ground. Falls are a frequent cause of mortality and morbidity and, often, limit autonomy leading to premature entry into assisted living facilities.

In Italy, in 2002 it was estimated that 28.6% of people over 65 years fall within a year: of these, 43% fall more than once and 60% of falls occur at home. Such falls can often result in fractures leading to the need for hospitalization with significant impact on both motor and cognitive function. Balance and gait rehabilitation are of primary importance for the recovery of a person's autonomy and independence, especially in older individuals who have undergone osteosynthesis or prosthesis surgery of the lower limbs. Technological and robotic rehabilitation allows for greater intensity, objectivity, and standardization in treatment protocols, as well as in outcome measurement. In this context, patient motivation is fuelled and maintained by both the sensory stimuli that support technological treatment and the challenge of achieving ever better results, objective feedback from instrumental assessments. Osteoarthritic patients who have undergone osteosynthesis or lower extremity prosthetic surgery require special attention, especially with the goal of preventing further accidents and reducing the patient's risk of falling.

Given these considerations, it is believed that conventional physical therapy combined with technological balance treatment may be more effective on rehabilitation outcome than conventional therapy alone.

DETAILED DESCRIPTION:
Twenty-four patients of both sexes will be recruited, evaluated, and treated at Rehabilitation and Physical Medicine Unit, Fondazione Policlinico Universitario A. Gemelli IRCCS of Rome, from August 2022 to August 2023. Patients will be divided into two groups by 1:1 randomization ratio: one group (Technological Group, TG) will perform specific rehabilitation for the balance using the robotic platform (Hunova®, Movendo Technology srl, Genova, IT) 3 times a week, for 4 weeks (12 total sessions), for 45 minutes of treatment, in addition to the conventional treatment and one group will perform only the conventional treatment (Control Group, CG), as per daily routine.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 55 years;
* Patients with outcomes of surgery for prosthetic hip or knee replacement;
* Latency from the acute event between 15 days and 3 months;
* Cognitive abilities to execute simple orders and understand the physical therapist's directions [assessed by Token Test (score ≥26.5)];
* Ability to walk independently or with little assistance;
* Ability to understand and sign informed consent.

Exclusion Criteria:

* Presence of systemic, neurological, cardiac pathologies that make walking hazardous or cause motor deficits;
* Presence of oncological pathologies;
* Presence of plantar ulcers;
* Partial or total amputation of foot segments.

Ages: 55 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale (BBS) | Change from Baseline Ambulation Index at 4 weeks
  The Berg Balance Scale (BBS) is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function and takes approximately 20 minutes to complete. It does not include the assessment of gait.

SECONDARY OUTCOMES:
Motricity Index (MI) | Change from Baseline Ambulation Index at 4 weeks
  The Motricity Index can be used to assess the motor impairment in a patient who has had a stroke. Test for each leg: (1) ankle dorsiflexion with foot in a plantar flexed position
  14 points are given if there is less than a full range of dorsiflexion (2) knee extension with the foot unsupported and the knee at 90° 14 points are given for less than 50% of full extension 19 points are given for full extension yet it can be easily pushed down (3) hip flexion with the hip bent at 90° moving the knee towards the chin 14 points are given if there is less than a full range of passive motion 19 points are given if the hip is fully flexed yet it can be easily pushed down. Interpretation: minimum score: 0 maximum score: 100
Timed Up and Go Test (TUG) | Change from Baseline Ambulation Index at 4 weeks
  The Timed Up and Go test (TUG) measures in seconds the time it takes a subject to rise from a chair, walk a distance of 3 meters, turn, walk back to the chair and sit down.
  The performance is rated on a scale of 1 to 5 (where 1 is normal and 5 is severely abnormal) according to the observer's perception of the patient's risk of falling.
  The timed part of the test records the mean time (in seconds) from initial getting up to re-seating. Patients are compared with the mean time of adults in their age group, 60 to 69, 70 to 79, and 80 to 99 years of age.
Knee Injury and Osteoarthritis Outcome Score - Italian Version (KOOS-I) | Change from Baseline Ambulation Index at 4 weeks
  KOOS-I is a self-administered questionnaire of 42 items and 5 sub-scales investigating different aspects: Symptoms (7 items, 2 inherent to stiffness); Pain (9 items); Functions and activities of daily living (17 items); Sports and recreation (5 items); and Quality of life in relation to the knee (4 items).
  All Scale Items present the same response mode by making use of a 5-point Likert scale ranging from 0 (no problems or difficulties) to 4 (high problems or difficulties).
Hip disability and Osteoarthritis Outcome Score - Italian version (HOOS-I) | Change from Baseline Ambulation Index at 4 weeks
  HOOS-I is a self-administered questionnaire designed to assess reported symptoms at the hip joint level in subjects with or without primary osteoarthritis and following hip arthroplasty surgery.
  HOOS-I consists of 40 items divided into 5 subscales that assess five distinct dimensions relevant to the patient: Symptoms (3 items on symptoms and 2 on stiffness); Pain (10 items); Activities of Daily Living (ADL) (17 items); Physical function, sports and leisure activities (4 items); Quality of life (4 items).
  The patient has to express his/her opinion through standardized response options based on the 5-point Likert scale (none, mild, moderate, severe, extreme); each response is assigned a score ranging from 0 (no problem) to 4 (extreme problems).
Ambulation Index (AI) | Change from Baseline Ambulation Index at 4 weeks
  The Ambulation Index is a rating scale to assess mobility by evaluating the time and degree of assistance required to walk 8 meters. Scores range from 0 (asymptomatic and fully active) to 10 (bedridden). The patient is asked to walk a marked 8 meters course as quickly and safely as possible. The examiner records the time and type of assistance (e.g., cane, walker, crutches) needed. Although the patient's walking is timed, the time is not used directly but is utilized in conjunction with other factors to rate the patient on an ordinal scale with 11 gradations.
  0 = Asymptomatic; fully active. 10 = Bedridden
Walking handicap scale (WHS) | Change from Baseline Walking handicap scale at 4 weeks
  The Walking handicap scale (WHS) is an assessment tool that allows us to evaluate the quality of walking in the home and social environment through a a scale comprising six categories.
  1 = Physiological walking: walking only as exercise 6 = Unrestricted walking in social settings: independent in all activities, on uneven ground, in crowded places, shows complete independence in public places
Functional Ambulation Classification (FAC) | Change from Baseline Functional Ambulation Classification at 4 weeks
  The Functional Ambulation Categories (FAC) is a functional walking test that evaluates ambulation ability. This 6-point scale assesses ambulation status by determining how much human support the patient requires when walking, regardless of whether or not they use a personal assistive device.
  To use the FAC, an assessor asks the subject various questions and briefly observes their walking ability to provide a rating from 0 to 5.
  A score of 0 indicates that the patient is a non-functional ambulator (cannot walk); A score of 1, 2 or 3 denotes a dependent ambulator who requires assistance from another person in the form of continuous manual contact (1), continuous or intermittent manual contact (2), or verbal supervision/guarding (3).
  A score of 4 or 5 describes an independent ambulator who can walk freely on: level surfaces only (4) or any surface (5=maximum score).
10 Meter Walk Test (10mWT) | Change from Baseline 10 Meter Walk Test at 4 weeks
  The 10mWT is used to assess walking speed in meters/second (m/s) over a short distance. The total time taken to ambulate 6 meters (m) is recorded to the nearest hundredth of a second. 6 m is then divided by the total time (in seconds) taken to ambulate and recorded in m/s.
  The time is measured for the middle 6 m to allow for patient acceleration and deceleration.
  The time is started when any part of the leading foot crosses the plane of the 2-m mark.
  The time is stopped when any part of the leading foot crosses the plane of the 8-m mark.1 The time to walk the middle 6m, the level of assistance, and type of assistive device and/or bracing used will be documented.
  If a patient requires total assistance or is unable to ambulate at all, a score of 0 m/s will be documented.
Six-Minute Walk test (6MWT) | Change from Baseline 10 Meter Walk Test at 4 weeks
  The six-minute walk test (6MWT) is a sub-maximal exercise test used to assess walking endurance and aerobic capacity. Participants will walk around the perimeter of a set circuit for a total of six minutes. The score of the test is the distance a patient walks in 6 minutes (measured in meters and can round to the nearest decimal point).
  Distance (in meters) covered in six minutes is calculated by multiplying the number of total laps by 12 meters and adding the distance of the partial lap completed at the time the test ended.
Modified Barthel Index (mBI) | Change from Baseline 10 Meter Walk Test at 4 weeks
  The modified Barthel Index (mBI) for activities of daily living is meant to be used in the assessment of patient performance (or degree of assistance required) with respect to self-care, sphincter management, transfers and locomotion. The index consist of 10 items (each scored with a number of points) that relate to activities of daily living (ADLs) where the final score is calculated by summing the points awarded to each item. A five-point rating scales for each item to improve sensitivity to detecting change.
  The 10 items assessed relate to help needed with feeding, bathing, grooming, dressing, transfers, walking, climbing stairs, presence or absence of fecal incontinence and urinary incontinence.
  The score ranges from 0 (maximum dependence) to 100 (maximum independence)
EuroQol- 5 Dimension (EQ-5D) | Change from Baseline 10 Meter Walk Test at 4 weeks
  EQ-5D is an instrument which evaluates the generic quality of life. The EQ-5D descriptive system is a preference-based HRQL measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The answers given to ED-5D permit to find 243 unique health states or can be converted into EQ- 5D index an utility scores anchored at 0 for death and 1 for perfect health.
Modified Fatigue Impact Scale (MFIS) | Change from Baseline 10 Meter Walk Test at 4 weeks
  The Modified Fatigue Impact Scale (MFIS) is an instrument that provides an assessment of the effects of fatigue in terms of physical, cognitive, and psychosocial functioning. The full-length MFIS consists of 21 items while the abbreviated version has 5 items.
  The MFIS is a structured, self-report questionnaire that the patient can generally complete with little or no intervention from an interviewer. However, patients with visual or upper extremity impairments may need to have the MFIS administered as an interview. Interviewers should be trained in basic interviewing skills and in the use of this instrument.
  The total score for the MFIS is the sum of the scores for the 21 items. Individual subscale scores for physical, cognitive, and psychosocial functioning can also be generated by calculating the sum of specific sets of items.
Fatigue Scale for Motor and Cognitive Function (FSMC) | Change from Baseline 10 Meter Walk Test at 4 weeks
  The FSMC is an assessment of MS-related cognitive and motor fatigue. A Likert-type 5-point scale (ranging from 'does not apply at all' to 'applies completely') produces a score between 1 and 5 for each scored question. Thus minimum value is 20 (no fatigue at all) and maximum value is 100 (severest grade of fatigue). Two subscales (mental and physical fatigue) can be made. Items included in the subscale mental are 1-4-7-8-11-13-15-17-18-20 and items included in the subscale physical are 2-3-5-6-9-10-12-14-16-19.
Frontal Assessment Battery (FAB) | Change from Baseline 10 Meter Walk Test at 4 weeks
  The FAB is a brief tool that can be used at the bedside or in a clinic setting to assist in discriminating between dementias with a frontal dysexecutive phenotype and Dementia of Alzheimer"s Type (DAT).
  The FAB has validity in distinguishing Fronto-temporal type dementia from DAT in mildly demented patients (MMSE > 24). Total score is from a maximum of 18, higher scores indicating better performance.
Trial Making Test (TMT) | Change from Baseline 10 Meter Walk Test at 4 weeks
  The Trail Making Test (TMT) measures flexibility of thinking on a visual-motor sequencing task. It consists of two parts, A and B, where 25 circles distributed over a sheet of paper. In Part A, the circles are numbered 1 - 25, and the patient should draw lines to connect the numbers in ascending order. In Part B, the circles include both numbers (1 - 13) and letters (A - L); as in Part A, the patient draws lines to connect the circles in an ascending pattern, but with the added task of alternating between the numbers and letters (i.e., 1-A-2-B-3-C, etc.).
  Results for both TMT A and B are reported as the number of seconds required to complete the task; therefore, higher scores reveal greater impairment.
  Trail A: Average 29 seconds, Deficient > 78 seconds, Rule of Thumb Most in 90 seconds Trail B: Average 75 seconds, Deficient > 273 seconds, Rule of Thumb Most in 3 minutes
Stroop Colour Word Test (SCWT) | Change from Baseline 10 Meter Walk Test at 4 weeks
  The Stroop Color and Word Test (SCWT) is a neuropsychological test extensively used to assess the ability to inhibit cognitive interference that occurs when the processing of a specific stimulus feature impedes the simultaneous processing of a second stimulus attribute, well-known as the Stroop Effect. The subject is asked to read the words in the first task, to name colors in the second and third tasks. It is necessary to mark both any mistakes made but also the time spent on each task. The cut-off for the error interference effect is 4.24, while the cut-off for the time interference effect is 36.92.
Cancellation Test of Digit (CTD) | Change from Baseline 10 Meter Walk Test at 4 weeks
  In the Cancellation Test of Digits (CTD) the patient is asked to cross out with a pencil, as quickly as possible, all numbers corresponding to those indicated at the top of each matrix. Line A serves as an example. The performance of the subject is counted from line I. Corrections of the barriers are not allowed. The task of the examiner is mark the point at which the subject has exceeded the maximum time of the test, but let the subject let the subject finish his task for each matrix. The maximum time for each matrix is 45 sec- and is considered from the moment the subject finishes the run in. If the subject takes less time than the maximum time, it will be indicated at the end of each matrix. The time cut-off for the test is 23.9.

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Giovannini, MD, phD, Principal Investigator — Fondazione Policlinico Universitaria A. Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] R Core Team (2021). R: A language and environment for statistical computing. R Foundation for Statistical Computing, Vienna, Austria. URL https://www.R-project.org/.
- [Result] Alessandri G, Zuffiano A, Perinelli E. Evaluating Intervention Programs with a Pretest-Posttest Design: A Structural Equation Modeling Approach. Front Psychol. 2017 Mar 2;8:223. doi: 10.3389/fpsyg.2017.00223. eCollection 2017. PMID 28303110
- [Result] Aprile I, Iacovelli C, Padua L, Galafate D, Criscuolo S, Gabbani D, Cruciani A, Germanotta M, Di Sipio E, De Pisi F, Franceschini M. Efficacy of Robotic-Assisted Gait Training in chronic stroke patients: Preliminary results of an Italian bi-centre study. NeuroRehabilitation. 2017;41(4):775-782. doi: 10.3233/NRE-172156. PMID 28946585
- [Result] Burnham KP, Anderson DR. Multimodel Inference: Understanding AIC and BIC in Model Selection. Sociological Methods & Research. 2004;33(2):261-304. doi:10.1177/0049124104268644
- [Result] Castelli L, De Luca F, Marchetti MR, Sellitto G, Fanelli F, Prosperini L. The dual task-cost of standing balance affects quality of life in mildly disabled MS people. Neurol Sci. 2016 May;37(5):673-9. doi: 10.1007/s10072-015-2456-y. Epub 2016 Jan 4. PMID 26728268
- [Result] Cattaneo D, Carpinella I, Aprile I, Prosperini L, Montesano A, Jonsdottir J. Comparison of upright balance in stroke, Parkinson and multiple sclerosis. Acta Neurol Scand. 2016 May;133(5):346-54. doi: 10.1111/ane.12466. Epub 2015 Aug 3. PMID 26234280
- [Result] Davis RB, Õunpuu S, Tyburski D, Gage JR. A gait analysis data collection and reduction technique. Hum. Mov. Sci. 1991; 10, 575-587
- [Result] Glyn-Jones S, Palmer AJ, Agricola R, Price AJ, Vincent TL, Weinans H, Carr AJ. Osteoarthritis. Lancet. 2015 Jul 25;386(9991):376-87. doi: 10.1016/S0140-6736(14)60802-3. Epub 2015 Mar 4. PMID 25748615
- [Result] Harris PA, Taylor R, Minor BL, Elliott V, Fernandez M, O'Neal L, McLeod L, Delacqua G, Delacqua F, Kirby J, Duda SN; REDCap Consortium. The REDCap consortium: Building an international community of software platform partners. J Biomed Inform. 2019 Jul;95:103208. doi: 10.1016/j.jbi.2019.103208. Epub 2019 May 9. PMID 31078660
- [Result] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Result] Hu LT, Bentler PM. Fit indices in covariance structure modeling: Sensitivity to underparameterized model misspecification. Psychological Methods. 1998, 3(4), 424-453. doi: 10.1037/1082-989X.3.4.424
- [Result] Hu LT, Bentler PM. Cutoff Criteria for Fit Indexes in Covariance Structure Analysis: Conventional Criteria versus New Alternatives. Structural Equation Modeling, 1999, 6, 1-55. doi: 10.1080/10705519909540118
- [Result] Julious, SA. 'Sample size of 12 per group rule of thumb for a pilot study'. Pharmaceutical Statistics. 2005, Vol 4. Pages 287-291.
- [Result] Kline, RB. (2016). Principles and Practice of Structural Equation Modeling, 4th Edn. New York, NY: The Guilford Press.
- [Result] MacCallum RC, Browne MW, Sugawara HM. Power analysis and determination of sample size for covariance structure modeling. Psychological Methods, 1996, 1(2), 130-149. doi: 10.1037/1082-989X.1.2.130
- [Result] Muthén, BO and Curran PJ. General longitudinal modeling of individual differences in experimental designs: a latent variable framework for analysis and power estimation. Psychol. Methods 1997, 2, 371-402. doi: 10.1037/1082-989X.2.4.371
- [Result] Prosperini L, Castelli L, De Luca F, Fabiano F, Ferrante I, De Giglio L. Task-dependent deterioration of balance underpinning cognitive-postural interference in MS. Neurology. 2016 Sep 13;87(11):1085-92. doi: 10.1212/WNL.0000000000003090. Epub 2016 Aug 12. PMID 27521436
- [Result] Prosperini L, Castelli L, Sellitto G, De Luca F, De Giglio L, Gurreri F, Pozzilli C. Investigating the phenomenon of "cognitive-motor interference" in multiple sclerosis by means of dual-task posturography. Gait Posture. 2015 Mar;41(3):780-5. doi: 10.1016/j.gaitpost.2015.02.002. Epub 2015 Feb 21. PMID 25770078
- [Result] Sinusas K. Osteoarthritis: diagnosis and treatment. Am Fam Physician. 2012 Jan 1;85(1):49-56. PMID 22230308